CLINICAL TRIAL: NCT03254654
Title: A Phase II, Single-center, Randomized Study of Vinorelbine Plus Apatinib Versus Vinorelbine as Second-Line or Third-Line Treatment in Patients With Advanced Triple-Negative Breast Cancer (NAN Trail)
Brief Title: Vinorelbine Plus Apatinib Versus Vinorelbine in Advanced Triple-Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xichun Hu, Vice Director of department of medical oncology, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fudan BR2017-23
Record Dates: First submitted 2017-08-17; First posted 2017-08-18 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Advanced Triple-Negative Breast Cancer
MeSH Terms: interventions — Vinorelbine; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vinorelbine Plus Apatinib (Experimental): Vinorelbine: 20 mg/m2, D6, D13, D20
  Apatinib: 250 mg/d, D1-5, D8-12, D15-19. The starting dose will be 250mg/d in the first cycle, if tolerable, 500 mg/d will be administered from the cycle 2.
  Interventions: Drug: Vinorelbine; Drug: Apatinib
- Vinorelbine (Active Comparator): Vinorelbine: 25 mg/m2, D1, D8, D15
  Interventions: Drug: Vinorelbine

INTERVENTIONS:
Drug: Vinorelbine — Experimental: 20 mg/m2, D6, D13, D20 Active Comparator: 25 mg/m2, D1, D8, D15
  Other Names: NVB
Drug: Apatinib — 250 mg/d, D1-5, D8-12, D15-19. The starting dose will be 250mg/d in the first cycle, if tolerable, 500 mg/d will be administered from the cycle 2.
  Arms: Vinorelbine Plus Apatinib

SUMMARY:
Vinorelbine Plus Apatinib Versus Vinorelbine in Advanced Triple-Negative Breast Cancer

DETAILED DESCRIPTION:
A Phase II, Single-center, Randomized Study of Vinorelbine Plus Apatinib Versus Vinorelbine as Second-Line or Third-Line Treatment in Patients With Advanced Triple-Negative Breast Cancer (NAN trail)

ELIGIBILITY:
Inclusion Criteria:

1. Performance Status 0-1
2. Life expectancy longer than 3 months
3. Histological proven unresectable recurrent or advanced breast cancer
4. Triple-negative for estrogen receptor (ER), progestogen receptor (PR), and human epithelial receptor-2 (HER2) by immunohistochemistry (ER <1%, PR <1% and Her2 negative). A negative Her2 gene amplification should be verified by FISH test for those patients with Her2 (2+)
5. Patients must have progressed after 1 or 2 prior chemotherapy regimens for metastatic disease, and consistent with the following treatment failure definition: progress in the first-line or second-line regimen treatment, or follow-up disease progression less than 3 months after completion of their last dose
6. At least one extracranial measurable disease according to the response evaluation criteria in solid tumor (RECIST 1.1)
7. Radiation therapy within 4 weeks prior to enrollment
8. All patients enrolled are required to have adequate hematologic, hepatic, and renal function
9. Be able to understand the study procedures and sign informed consent

Exclusion Criteria:

1. Patients had prior treatment with vinorelbine
2. Pregnant or lactating women, women of child-bearing potential, unwilling to use adequate contraceptive protection during the process of the study
3. Patients with symptomatic central nervous system metastases are not permitted, except for those with stable and asymptomatic brain metastases who have completed cranial irradiation, and have at least one measurable lesion outside the brain. Radiotherapy should be completed within 4 weeks prior to the registration
4. Treatment with an investigational product within 4 weeks before the first treatment
5. Severe cardiopulmonary insufficiency, severe hepatic and renal dysfunction
6. Uncontrolled serious infection
7. Unhealed wound or bone fracture
8. Patients with hypertension and uncontrolled hypertension with hypotensive drugs therapy (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg). Patients with grade I or above myocardial ischemia or myocardial infarction or arrhythmia (including QT interval ≥ 440 ms) or cardiac insufficiency
9. Inability to swallow, gastrointestinal resection, chronic diarrhea and obstruction of the intestine, various factors which affect drug use and absorption
10. Coagulation disorders (PT > 16 s, APTT > 43 s, TT > 21 s, Fbg < 2g / L) Being treated with thrombolytic or anticoagulant therapy, with bleeding tendency or definite gastrointestinal bleeding concerns (eg: local active ulcer lesions, fecal occult blood + + or above)
11. Artery or venous thrombosis occurred within 6 months before the study begins, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis, and pulmonary embolism, etc.
12. Patient who has a history of psychotropic substance abuse and is unable to stop or have a history of mental disorders
13. Have received prior treatment with a VEGFR TKI (Bevacizumab is permitted)
14. Another malignancy within 5 years, except for cured basal cell carcinoma of the skin and cervical carcinoma

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
PFS | 6 weeks
  Progression Free Survival

SECONDARY OUTCOMES:
OS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Overall Survival
ORR | 6 weeks
  Objective Response Rate
Safety: Number of Participants with Adverse Events | 6 weeks
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, China